CLINICAL TRIAL: NCT05144061
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) of HRS2398 in Subjects With Advanced Malignant Tumors
Brief Title: A First-in-human Study of HRS2398 Tablets in Subjects With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS2398-I-101
Record Dates: First submitted 2021-10-12; First posted 2021-12-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2022-11

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Intervention Model Description: Single therapy of HRS2398
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): HRS2398 Tablets
  Interventions: Drug: HRS2398 Tablets

INTERVENTIONS:
Drug: HRS2398 Tablets — Take 5mg to 320mg once or twice a day ; Oral administration , 21 days as a cycle.

SUMMARY:
The study is being conducted to determine the dose limited toxicity(DLT) and maximum tolerated dose(MTD) and recommended Phase 2 dose(RP2D) of HRS2398 in subjects with advanced malignant tumor ; The second objectives is to evaluate safety and preliminary efficacy and PK profile of HRS2398 in subjects with advanced malignant tumor ; Exploratory cohort is to explore the relationship between gene mutation and efficacy and resistance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. subjects ≥18 years and ≤70 years.
3. Patients with Histologically or cytologically confirmed advanced Malignant tumors who had failed standard treatment or had not been treated with standard therapy.
4. ECOG ≤1.
5. Subjects with life expectancy of ≥ 3 months.
6. At least one measurable lesion ( RECIST version 1.1).
7. Subjects must have adequate organ function (whole blood or component transfusion or BFGF within 2 weeks before 1st dose of study drug is prohibited):

   1. Absolute neutrophil count (ANC) ≥1.5 x10^9/L;
   2. Platelet count ≥ 100 x 10^9/L;
   3. Hemoglobin ≥ 90 g / L;
   4. Total bilirubin (TBil) ≤1.5 x ULN;
   5. Liver function tests alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN, for patients with known liver cancer or liver metastases, AST and ALT ≤ 5 x ULN;
   6. Gr ≤ 1.5x ULN or an estimated glomerular filtration rate (eGFR) > 50 mL/min;
   7. INR ≤1.5 x ULN and APTT ≤ 1.5 x ULN;
   8. LVEF≥50%，QTc Male: <450ms; Female: <470ms.
8. Subjects (males and females) of childbearing potential should be willing to use reliable contraception methods that are deemed effective by the investigator from visit 1 through 180 days following the last dose of study drug.
9. Archived wax lump tumor tissue samples or biopsy and blood sample collection during screening period.
10. As judged by the investigator, can follow protocol.

Exclusion Criteria:

1. Untreated and/or uncontrolled brain metastases.
2. Patients with clinical symptoms of cancer ascites, pleural effusion, who need to drainage, or who have undergone ascites drainage within 2 weeks prior to the first administration.
3. Failure to recover from adverse events from the most recent anti-tumor treatment to CTCAE ≤ grade2.
4. Inability to swallow tablets or gastrointestinal disease, possible impairment of adequate absorption of study drugs.
5. Have severe cardiac disease:NYHA class ≥grade II heart failure; unstable angina pectoris；myocardial infarction within 12 months； clinically significant supraventricular or ventricular arrhythmias require treatment or intervention; Hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
6. Known active hepatitis C virus, or known active hepatitis B virus.
7. Allergic to the HRS2398 or the similar drug.
8. Concurrent anticancer treatment or use of other investigational product within 4 weeks before start of trial treatment; major surgery, radiotherapy, chemotherapy within 4 weeks before 1st dose of trial treatment.
9. The patient is currently using a drug known to be a strong inhibitor of CYP3A4 within 2 weeks before 1st dose of study drug ，or strong inducer of CYP3A4 within 4 weeks before 1st dose of study drug .
10. The investigator determined that the patient should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | up to 21 days
Maximum tolerated dose（MTD） | up to 6 months
Recommended Phase II Dose (RP2D) | up to 21 days

SECONDARY OUTCOMES:
Number of subjects with adverse events and the severity of adverse events | from the first drug administration to within 30 days for the last treatment dose
Cmax of HRS2398 of Single administration | Single administration : 30min before administration of Day1, 5min, 0.25 hour, 0.5 hour, 0.75 hour, 1 hour , 2hours, 4hours, 6hours, 8hours, 10hours, 24hours, 48hours, 72hours after administration of Day1
Tmax of HRS2398 of Single administration | Single administration : 30min before administration of Day1, 5min, 0.25 hour, 0.5 hour, 0.75 hour, 1 hour , 2hours, 4hours, 6hours, 8hours, 10hours, 24hours, 48hours, 72hours after administration of Day1
AUC0-t of HRS2398 of Single administration | ingle administration : 30min before administration of Day1, 5min, 0.25 hour, 0.5 hour, 0.75 hour, 1 hour , 2hours, 4hours, 6hours, 8hours, 10hours, 24hours, 48hours, 72hours after administration of Day1
AUC0-12 of HRS2398 of Single administration | Single administration : 30min before administration of Day1, 5min, 0.25 hour, 0.5 hour, 0.75 hour, 1 hour , 2hours, 4hours, 6hours, 8hours, 10hours after administration of Day1
T1/2 of HRS2398 of Single administration | Single administration : 30min before administration of Day1, 5min, 0.25 hour, 0.5 hour, 0.75 hour, 1 hour , 2hours, 4hours, 6hours, 8hours, 10hours, 24hours, 48hours, 72hours after administration of Day1
Cmax of HRS2398 of Multiple doses | Multiple administration: Day8, Day15, Day17 of Cycle1, Day1 of Cycle2-4 (each cycle is 21 days)
Tmax of HRS2398 of Multiple administration | Multiple administration: Day8, Day15, Day17 of Cycle1, Day1 of Cycle2-4 (each cycle is 21 days)
AUC0-t of HRS2398 of Multiple administration | Multiple administration: Day8, Day15, Day17 of Cycle1, Day1 of Cycle2-4 (each cycle is 21 days)
AUC0-12 of HRS2398 of Multiple administration | Multiple administration: Day8, Day15, Day17 of Cycle1, Day1 of Cycle2-4 (each cycle is 21 days)
T1/2 of HRS2398 of Multiple administration | Multiple administration: Day8, Day15, Day17 of Cycle1, Day1 of Cycle2-4 (each cycle is 21 days)
Bioavailability of fasting state | up to 4 months
  PK blood samples from subjects were collected for bioavailability ，Postprandial AUC divided by fasting AUC
Objective Response Rate(ORR) | up to 4 months
  Radiological scans performed at baseline then every 6 weeks until objective radiological disease progression
Disease Control Rate(DCR) | up to 4 months
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST 1.1
Duration of response (DoR) | up to 4 months
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response
Progression free survival(PFS) | up to 4 months
  Defined as Progression free survival per RECIST 1.1 criteria according to Investigator's assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University/Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided